CLINICAL TRIAL: NCT03771391
Title: Multicentre Study Project to Evaluate the New Generation of Protein Supplements With Glycomacropeptide (GMP) in Patients With Phenylketonuria (PKU) Aged 10 Years and Older Over a 16 Week Period.
Brief Title: A 16 Week Study Evaluating the Introduction of a GMP Based Protein Substitute in Participants With PKU
Acronym: GMP In PKU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Collaborators: Kreiskliniken Reutlingen (Other); Johannes Gutenberg University Mainz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MCT-W-PKUSp-2017-06-29; F-2018-043 (Other: Landesärztekammer Baden-Württemberg)
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Phenylketonurias
Keywords: Phenylketonuria; PKU; Child; Children; Adult; Adults; GMP; Glycomacropeptide; Amino acid mixture; Amino acid; Protein supplement; Protein substitute
MeSH Terms: conditions — Phenylketonurias | interventions — caseinomacropeptide

STUDY DESIGN:
Intervention Model Description: The study has a stepped wedge design, which is chosen over the alternative cross-over study as it allows that all participants start on the amino acid supplement and avoids the difficulty of the 'wash-out' period being the same as one of the treatment strategies being offered.
Who Masked: Participant
Masking Description: At the point of randomisation every effort will be made to ensure that participants are unaware of the cluster they are randomised to; this is to help ensure that compliance is not affected by participants knowing when they will start the new treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4 Weeks (Experimental): All patients randomised to this arm will start on an amino acid based protein substitute and they will all swtich over to incorprating PKU Sphere after 4 weeks.
  Interventions: Dietary Supplement: PKU Sphere
- 8 Weeks (Experimental): All patients randomised to this arm will start on an amino acid based protein substitute and they will all swtich over to incorprating PKU Sphere after 8 weeks.
  Interventions: Dietary Supplement: PKU Sphere
- 12 Weeks (Experimental): All patients randomised to this arm will start on an amino acid based protein substitute and they will all swtich over to incorprating PKU Sphere after 12 weeks.
  Interventions: Dietary Supplement: PKU Sphere

INTERVENTIONS:
Dietary Supplement: PKU Sphere — PKU sphere is a powdered, low phenylalanine protein substitute containing a balanced mix of casein glycomacropeptide (GMP) isolate, essential and non-essential amino acids, carbohydrate, vitamins, minerals and docosahexaenoic acid (DHA). With sugar and sweetener.
  Other Names: GMP; Glycomacropeptide

SUMMARY:
This study aims to measure changes in participants' blood phenylalanine (Phe) levels in participants with PKU when switching from a conventional amino acid based protein substitute to a GMP based protein substitute (PKU Sphere) over a 16 week period.

DETAILED DESCRIPTION:
This is a stepped wedge, open-label study of PKU Sphere for the dietary management of participants with Phenylketonuria. It will be carried out with 33 participants who will be randomised into one of three clusters. The total study length per patient is 16 weeks. Each cluster transitions from taking their standard amino acid product alone to incorporating PKU Sphere (at least 50% of their protein substitue requirement) at different timepoints: week 5, 9 or 13.

Participants will have a face-to-face clinical review at the time of recruitment (week 0) and at 16 weeks (completion of the study). They will also have an additional telephone review when they switch onto PKU Sphere.

Blood samples will be taken at baseline, and then every two weeks for the duration of the study.

In addition to these study visits and procedures, routine clinical care will continue in line with local guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU made in neonatal period
* Treated by a low-phenylalanine diet and necessity of intake of at least one protein substitute per day
* Aged 10 years and above
* Three blood Phe measurements taken within the preceding six months
* Willing to replace current amino acid based protein substitute with PKU Sphere
* Ability to take at least 50% of protein requirements as PKU Sphere
* Ability to comply with the study protocol, in the opinion of the investigator
* Willingly given, written, informed consent from patient or parent/guardian
* Willingly given, written assent (if appropriate)

Exclusion Criteria:

* Women who are pregnant or planning to become pregnant during the study period
* Participants with atypical PKU (e.g. BH4 deficient)
* Intake of sapropterin dihydrochloride (Kuvan) in the six weeks prior to recruitment in the study
* Patients with soya, milk or fish allergies
* Any other severe disease

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change in blood Phe | Baseline (week 0) and weeks 2, 4, 6, 8, 10, 12, 14 and 16.
  Change in blood Phe concentrations when switching from an amino acid based protein substitute to a GMP based one (PKU Sphere). A minimum of five (5) blood samples (including a baseline measurement and one from each treatment arm) will be required for a patient to be included in the final analysis.

SECONDARY OUTCOMES:
Change in blood tyrosine | Baseline (week 0) and weeks 2, 4, 6, 8, 10, 12, 14 and 16.
  Impact of a GMP based protein substitute on blood tyrosine levels. A minimum of five (5) blood samples (including a baseline measurement and one from each treatment arm) will be required for a patient to be included in the final analysis.
Dietary intake | Weeks 1 and 16.
  Compliance with a low protein diet - 3-day food diary.
Protein substitute intake | Weeks 1, 4, 8, 12 and 16
  Compliance with the recommended volume of protein substitute - 3-day protein substitute diary.
Stool patterns | Weeks 1, 4, 8, 12 and 16
  3-day diary noting stool type (Bristol stool chart).
Satiety questionnaire | Weeks 1, 4, 8, 12 and 16
  Short questionnaire asking participants to consider their satiety levels over the last 7 days, asking them if it has increased, stayed the same or decreased. Questionnaire validated as part of a bachelor thesis.
Acceptance questionnaire | Weeks 1, 4, 8, 12 and 16
  Questionnaire to collect information about taste, odour and practicability of the protein substitutes. The questions are answered on a scale of 1 (bad) to 5 or 6 (good). Questionnaire validated as part of a bachelor thesis.
Gastrointestinal symptoms questionnaire | Weeks 1, 4, 8, 12 and 16
  Short questionnaire asking participants to consider their general gastrointestinal health over the previous 7 days. The occurrence of various GI symptoms are given as never, rare, often or always. Questionnaire validated as part of a bachelor thesis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Freisinger, Principal Investigator — Kreiskliniken Reutlingen GmbH
Locations (1):
- Kreiskliniken Reutlingen, Reutlingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No